CLINICAL TRIAL: NCT02330796
Title: A RANDOMIZED, MULTICENTRE PHASE IIa OPEN-LABEL, ACTIVE-COMPARATOR TRIAL TO ASSESS THE EFFICACY AND SAFETY OF TWO REGIMENS OF BUCILLAMINE 100 MG TABLETS AS COMPARED TO COLCHICINE 0.6 MG TABLETS FOR THE TREATMENT OF AN ACUTE GOUT FLARE IN SUBJECTS WITH MODERATE TO SEVERE GOUT.
Brief Title: Bucillamine for the Treatment of Acute Gout Flare in Subjects With Moderate to Severe Gout
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Revive Therapeutics, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: REV-201
Record Dates: First submitted 2014-12-31; First posted 2015-01-05 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-10

CONDITIONS: Gout
MeSH Terms: conditions — Gout | interventions — bucillamine; Colchicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm A (Experimental): Bucillamine (900 mg total dose over 7 days)
  Interventions: Drug: Bucillamine
- Arm B (Experimental): Bucillamine (1,800 mg total dose over 7 days)
  Interventions: Drug: Bucillamine
- Arm C (Active Comparator): Colchicine (1.8 mg total dose in 2 doses taken 1 hour apart)
  Interventions: Drug: Colchicine

INTERVENTIONS:
Drug: Bucillamine — Bucillamine Tablets
  Arms: Arm A; Arm B
Drug: Colchicine
  Arms: Arm C

SUMMARY:
A Phase IIA, open-label, multicenter, active-controlled, parallel-group clinical trial designed to evaluate the safety and efficacy of two doses of Bucillamine compared with low-dose Colchicine in the treatment of patients with acute gout flare.

DETAILED DESCRIPTION:
To evaluate the safety and tolerability of two regimens of Bucillamine 100 mg (900 mg and 1,800 mg) over seven days of treatment compared with Colchicine 0.6 mg (1.8 mg) in the treatment of patients with acute gout flare

ELIGIBILITY:
Inclusion Criteria:

* Subjects must present with confirmed diagnosis of gout, meeting the American College of Rheumatology (ACR) 1977 preliminary criteria for the classification of acute arthritis of primary gout
* Subjects must have experienced at least one (1) acute gouty arthritic attack in the 12 months prior to randomization
* Presence of acute gout flare for no longer than 3 days at Visit 2
* Pain intensity at inclusion (Visit 2) of 7-10 on 11-point PI-NRS (defined as severe gout flare for this study)
* All patients should not have contraindications for Colchicine use
* Subjects with a history of intolerance to NSAIDs (Checklists Checklist 1)
* Subjects with significant medical contraindication to NSAIDs (Checklist 2)
* Subjects with past failure of NSAIDs to control acute gouty arthritis attacks in the previous 12 months (Checklist 3)
* Regarding significant medical contraindication to NSAIDs or past failure of NSAIDs to control acute gouty arthritis attacks in the previous 12 months (i.e. refractoriness to NSAIDs) the patient must meet one of below criteria:

  1. At least one historical episode within the previous 12 months of being refractory or intolerant to NSAIDs that makes the physician concerned to use NSAIDs for a subsequent acute gout attack
  2. The current (referring) physician judgment is that NSAIDs are not appropriate for treating the patient's gouty arthritis flare which may be due to changes in patient status such as worsening co-morbid conditions or co-medications (e.g., GI tract disease, renal insufficiency, hypertension, fluid retention, concurrent use of diuretics and/or an angiotensin converting enzyme inhibitor or angiotensin receptor blocker, especially in CKD)
* Subjects must be willing and able to give written informed consent. A HIPAA and/or state privacy consent must also be signed
* Subjects must be able to swallow tablets
* Use of permitted concomitant medications must be unchanged in dose and or frequency, 30 days prior to screening
* Adequate organ function, evidenced by the following laboratory results within 90 days prior to randomization (historical lab results are acceptable).
* Creatine clearance > 45 mL/min based on Cockroft-Gault glomerular filtration rate (GFR) estimation
* For women of childbearing potential and men with partners of childbearing potential, agreement to use a highly effective, non-hormonal form of conception.

Exclusion Criteria:

* Subjects with rheumatoid arthritis, psoriatic arthritis, evidence/suspicion of infectious/septic arthritis, acute polyarticular gout (4 or more joints), with arthritis due to any cause other than gout that may confound any study assessments per Investigator discretion
* Subjects who have experienced >2 acute gouty arthritic attacks per month, or >12 attacks overall, in the 6 months prior to randomization
* Subjects with a history of myocardial infarction, unstable angina, cerebrovascular events, or coronary artery bypass grafting within the previous 6 months prior to screening
* Subjects with a Body Mass Index >45 kg/m2; calculated as body weight (kg)/height (m)2 at Screening Visit
* Subjects with acute or chronic infections including known HIV and/or Hepatitis B or C
* Uncontrolled hypertension (>160/90 mmHg seated) (if the first set of BP assessment meets the definition of uncontrolled hypertension, a second set of BP assessments may be performed after the patient has rested for at least 30 min. If the second set of BP assessments does not meet the definition of uncontrolled hypertension the patient will be eligible for participation)
* Subjects with proteinuria ≥1+ or ≥30 mg on dipstick urinalysis that is confirmed on repeat assessment within 24 hours
* Subjects with significant heart failure and activity impairment (Class III-IV of the New York Heart Association (NYHA)
* Subjects with any history of malignancy, 5 years prior to randomization
* Subjects with CKD NKF stages 3B -5 chronic renal dysfunction (eGFR <45 mL/min/1.73m2 acc. to Cockcroft Gault formula)
* Subjects with serious hepatic disorder (Child-Pugh scores B or C)
* Subjects who have not washed out of dopamine antagonists or depleting drugs excluding anticholinergics and/or antihistamines with anticholinergic effects at least 14 days prior to Day 1 (Visit 2)
* Subjects with a documented history of alcohol or substance abuse within the 12 months prior to randomization(consumption of >21 units of alcohol per week is considered alcohol abuse)
* Subjects with significant CNS effects including vertigo and dizziness

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2015-04; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Composite measure of adverse events (AEs), physical examinations, electrocardiograms (ECGs), vital signs, clinical laboratory evaluations, medical history, and prior/concomitant medications | 7 days
At least a 50% reduction in target joint pain PI-NRS score from baseline without using rescue drug | 72 hours

SECONDARY OUTCOMES:
A greater than or equal to 50% reduction in target joint pain PI-NRS score from baseline at 24 hours and 48 hours post-dose without using rescue drug | 24 hrs and 48 hrs

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - West Coast Research, San Roman, California
  - Texas Physicians Research Medical Group, Arlington, Texas
  - Sun Research Institute, San Antonio, Texas